CLINICAL TRIAL: NCT01018992
Title: Evaluation of the Efficacy of the CRF1 Antagonist GSK561679 in Women With Post-traumatic Stress Disorder
Brief Title: Evaluation of GSK561679 in Women With Post-Traumatic Stress Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Boadie W. Dunlop, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: IRB00022717; MH069056 (Other: Other)
Record Dates: First submitted 2009-11-06; First posted 2009-11-25 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-01

CONDITIONS: Stress Disorders, Post-Traumatic
Keywords: PTSD; Anxiety Disorder; Corticotropin releasing factor; Women
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders | interventions — NBI 77860; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Adult women with DSM-IV defined PTSD will receive matching placebo for 6 weeks
  Interventions: Drug: Placebo
- GSK561679 (Experimental): Adult women with DSM-IV-defined PTSD will receive GSK561679 at a fixed dose of 350 mg/day for 6-weeks
  Interventions: Drug: GSK561679

INTERVENTIONS:
Drug: GSK561679 — GSK561679, oral administration, 350mg/day, 6 week administration
  Other Names: CRF1 antagonist
  Arms: GSK561679
Drug: Placebo — Matching placebo, oral administration, 1 pill/day for 6 weeks
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
This study will test the hypothesis of whether an antagonist at the corticotropin releasing factor type 1 (CRF1) receptor (i.e. GSK561679) is superior to placebo in reducing symptoms of post-traumatic stress disorder (PTSD).

DETAILED DESCRIPTION:
Post-traumatic stress disorder (PTSD) is a chronic and common anxiety disorder that follows exposure to an overwhelming traumatic event. The majority of patients with PTSD also meet criteria for other psychiatric disorders and PTSD is associated with an increased risk for suicide attempts.

PTSD is responsive to psychological and pharmacological treatments, such as selective serotonin reuptake inhibitors (SSRIs), but response rates rarely exceed 60%, and even fewer patients (20-30%) achieve clinical remission. Thus, there is a clear need to develop novel and improved therapeutics for PTSD.

The study is divided into 4 phases:

Phase 1 (Screening): a 1 week no drug screening period to assess study eligibility.

Phase 2 (Pre-Treatment Testing Period): Eligible patients will be enrolled into a 1 week Testing Phase, which will include neuropsychological and neurophysiological testing as well as blood draws and electrocardiogram.

Phase 3 (Treatment Period): Eligible patients will be enrolled in a two-armed 6-week period of double-blind placebo-controlled acute treatment. All subjects who continue to meet eligibility criteria will be randomized to one of two groups: GSK561679 (at a fixed dose of 350 mg/day) or placebo. Randomization will be performed at a 1:1 ratio into two treatment groups. Neuropsychological and neurophysiological testing will be repeated after 5 weeks of the double-blind treatment period.

Phase 4 (Follow-up Period): Safety follow-up visits will be conducted 1 week and 1 month after the end of the treatment Phase 3.

ELIGIBILITY:
Inclusion Criteria:

* Female between 21-65 years of age
* Able to provide consent and willing to participate in research
* Fulfills Diagnostic and Statistical Manual of Mental Disorders, 4th edition (DSM-IV) criteria for primary diagnosis of PTSD
* PTSD duration of illness at least 3 months
* Able to provide consent and willing to participate in research
* CAPS score of ≥ 50 at Screening and Visit 3 (randomization)
* Negative Urine toxicology test
* Agrees to use protocol-defined effective birth control method
* If the patient has a history of peptic ulcer disease (PUD), there is documentation of the etiology of the PUD and that effective treatment was provided with full eradication of ulcers and symptoms

Exclusion Criteria:

* Lifetime or current diagnosis of schizophrenia or other psychotic disorder, bipolar disorder, obsessive compulsive disorder (OCD), or current Axis I disorder [(except for major depression secondary to the PTSD, dysthymia, depression not otherwise specified (NOS) and anxiety disorders (panic disorder, social phobia, generalized anxiety disorder (GAD), specific phobia)]
* Subject is currently participating in another clinical trial in which she is or will be exposed to an investigational or non-investigational drug or device, or has done so within the preceding month for studies unrelated to PTSD, or 1 month for studies related to PTSD
* Current evidence or history of significant unstable medical illness or organic brain impairment, including stroke, central nervous system (CNS) tumor, demyelinating disease, cardiac, pulmonary, gastrointestinal, renal or hepatic impairment that would likely interfere with the action, absorption, distribution, metabolism, or excretion of GSK561679.
* Patients who in the investigator's judgment pose a current suicidal or homicidal risk
* DSM-IV substance abuse or dependence within the past 90 days. Subject has a positive test for illegal substances.
* Diagnosis of anorexia nervosa or bulimia in the past year.
* Subject has a documented history of hepato-biliary disease including a history of, or positive laboratory results for hepatitis (hepatitis B surface antigen and/or hepatitis C antibody), and/or clinically significant hepatic enzyme elevation including any one of the following enzymes greater than 1.5 times the upper limit of normal (ULN) value (alanine transaminase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), total or direct bilirubin > 1.5 x ULN, unless consistent with presumed or diagnosed Gilbert's disease)
* Subject has taken systemic corticosteroids within 2 weeks of the Randomization Visit
* Treatment with any other psychoactive medication within 2 weeks of Visit 1, including all antidepressants, psychoactive herbal or nutritional treatment (St Johns Wort, SAM-e), lithium, other mood stabilizers, oral antipsychotics, depot antipsychotics within 12 weeks, beta blockers, thioridazine, pimozide, opiates, anxiolytics, and sedatives (with the exception of zolpidem, eszopiclone, and zaleplon). Also any treatment with any medication that the PI judges not acceptable for this study.
* Subject who is likely to require the use of the following medications: Chronic (for more than 2 weeks), regular nonsteroidal anti-inflammatory drugs (NSAID) use. Any use of aspirin (including low dose)
* Subject has taken non-psychoactive (prescription or non-prescription), dietary, or herbal products, with a narrow therapeutic index, that are metabolized via the cytochrome P450 3A4 or 2C9 pathway (warfarin), or transported via OATP1B1 or P-gp, within 2 weeks (or 5 half-lives, whichever is longer) prior to the Randomization Visit.
* Subject has taken other (non-psychoactive) prescription, non-prescription, dietary, or herbal products that are potent inducers or inhibitors of the cytochrome P450 3A4 pathway for 2 weeks (or 5 half lives, whichever is longer) prior to the Randomization Visit.
* Subject has a stool positive for occult blood.
* Pregnancy or lactation
* Subjects who, in the opinion of the investigator, would be non compliant with the visit schedule or study procedures (e.g. illiteracy, planned vacations, or planned hospitalizations during the study).
* Previous treatment with CRF1 receptor antagonist
* Any laboratory abnormality that in the investigator's judgment is considered to be clinically significant (blood pressure, electrocardiogram (ECG), thyroid stimulating hormone (TSH), liver function test (LFT), etc.)
* Patients who are receiving exposure-based psychotherapy that targets PTSD symptoms
* Current or planned litigation or other actions related to secondary gain regarding the traumatic event
* Subject has clinical evidence of, or ECG results indicating any of the following at either screen or Randomization Visit unless repeat ECG shows that the parameter had returned to within normal range by the Randomization Visit:

  1. Corrected QT Interval (QTc) > 450 msec;
  2. any cardiac condition or ECG evidence that the investigator feels may predispose the subject to ischemia or arrhythmia; or
  3. any ECG abnormality that, in the investigator's judgment, may pose a potential safety concern

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2009-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boadie Dunlop, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Stress and Health Research Program, San Francisco VA Medical Center, University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia
  - Mount Sinai School of Medicine, New York, New York
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Derived] Jovanovic T, Duncan EJ, Kaye J, Garza K, Norrholm SD, Inslicht SS, Neylan TC, Mathew SJ, Iosifescu D, Rothbaum BO, Mayberg HS, Dunlop BW. Psychophysiological treatment outcomes: Corticotropin-releasing factor type 1 receptor antagonist increases inhibition of fear-potentiated startle in PTSD patients. Psychophysiology. 2020 Jan;57(1):e13356. doi: 10.1111/psyp.13356. Epub 2019 Feb 26. PMID 30807663
- [Derived] Pape JC, Carrillo-Roa T, Rothbaum BO, Nemeroff CB, Czamara D, Zannas AS, Iosifescu D, Mathew SJ, Neylan TC, Mayberg HS, Dunlop BW, Binder EB. DNA methylation levels are associated with CRF1 receptor antagonist treatment outcome in women with post-traumatic stress disorder. Clin Epigenetics. 2018 Nov 3;10(1):136. doi: 10.1186/s13148-018-0569-x. PMID 30390684
- [Derived] Dunlop BW, Rothbaum BO, Binder EB, Duncan E, Harvey PD, Jovanovic T, Kelley ME, Kinkead B, Kutner M, Iosifescu DV, Mathew SJ, Neylan TC, Kilts CD, Nemeroff CB, Mayberg HS. Evaluation of a corticotropin releasing hormone type 1 receptor antagonist in women with posttraumatic stress disorder: study protocol for a randomized controlled trial. Trials. 2014 Jun 21;15:240. doi: 10.1186/1745-6215-15-240. PMID 24950747

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Emory University School of Medicine, Mount Sinai School of Medicine, Baylor College of Medicine, and the University of California San Francisco between January 2010 and June 2014.
Pre-assignment Details: Subjects stopped psychotropic medications (w/ the exception of zolpidem, eszopiclone, and zaleplon for insomnia) w/in 2 weeks (6 weeks for fluoxetine) of Visit 1. Patients on ineffective psychotropic medications tapered off by the patients' prescribing doctor. 139 subjects did not proceed to randomization due to meeting exclusionary criteria.
Groups:
- GSK561679: Adult women with DSM-IV-defined PTSD received GSK561679 at a fixed dose of 350 mg/day for 6-weeks
- Placebo: Adult women with DSM-IV defined PTSD received matching placebo for 6 weeks
Period: Overall Study
Arm/Group | GSK561679 | Placebo
Started | 63 | 65
Completed | 47 | 49
Not Completed | 16 | 16
Not completed — Adverse Event | 8 | 3
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Protocol Violation | 0 | 4
Not completed — Lost to Follow-up | 5 | 1

BASELINE CHARACTERISTICS:
Population: All participants randomized to receive the double-blind study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK561679 | Placebo | Total
Number analyzed (Participants) | 63 | 65 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 65 | 128
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 65 | 128
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Efficacy, Measured by Change in the Clinician-Administered PTSD Scale (CAPS) Score
Description: The CAPS is a semi-structured clinical interview providing a measure of the severity of PTSD symptoms. A severity score is calculated by summing the frequency and intensity scores for each of the 17 DSM-IV criteria symptoms. The severity of symptoms is rated on a scale from 0-4, where, 0 = Absent, 1 = Mild/subthreshold; 2 = Moderate/ threshold, 3 = Severe/markedly elevated and 4 = Extreme/ incapacitating. Scores may range from 0 (no symptoms) to 136 (severe symptoms). Change is the difference in scores between baseline and 6 weeks.
Time Frame: Baseline, Week 6
Population: Intent to treat analysis was performed using maximum likelihood estimation with mixed models to include all observations.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
Score on a scale | -26.02 (22.28) | -27.33 (19.76)

2. Secondary Outcome: Efficacy, Measured by Response Rate of at Least 50% Improvement in CAPS Score at the End of 6 Weeks as Compared to Baseline
Description: The number of participants that showed at least a 50% reduction in CAPS scores from their baseline visit at the end of 6 weeks were measured has having a response to the treatment. The CAPS is a semi-structured clinical interview providing a measure of the severity of PTSD symptoms. A severity score is calculated by summing the frequency and intensity scores for each of the 17 DSM-IV criteria symptoms. Scores may range from 0 (no symptoms) to 136 (severe symptoms).
Time Frame: Baseline, Week 6
Population: Intent to treat analysis was performed with missing subjects considered to be non-responders.
Measure: Number; unit: participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
participants | 14 | 18

3. Secondary Outcome: Efficacy, Measured by Change in the Montgomery-Asberg Depression Rating Scale (MADRS) Score
Description: The MADRS is a ten-item clinician-administered questionnaire used to measure the severity of depressive symptoms in patients with depressive disorders. Higher MADRS score indicates more severe depression, and each item yields a score of 0 to 6. The overall score ranges from 0 to 60. Change is the difference in scores between baseline and 6 weeks.
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
Score on a scale | -7.83 (9.32) | -5.98 (9.10)

4. Secondary Outcome: Safety, Measured by the Number of Subjects That Experienced an Adverse Event
Description: The occurrence of adverse events will be recorded at the end of 6 weeks.
Time Frame: Week 6
Population: Intent to Treat
Measure: Number; unit: participants
Arm/Group | GSK561679 | Placebo
Number analyzed (Participants) | 63 | 65
participants | 55 | 55

ADVERSE EVENTS:
Arm/Group | GSK561679 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/63 | 1/65
Other Adverse Events (participants affected / at risk) | 55/63 | 55/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | GSK561679 (N=63) | Placebo (N=65)
Asthma exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anaphylaxis (Immune system disorders) | 0 | 1 — Anaphylactic reaction to seafood in person with known allergy to seafood
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | GSK561679 (N=63) | Placebo (N=65)
Headache (Nervous system disorders) | 25 | 24
Nausea (Gastrointestinal disorders) | 19 | 11
Insomnia (Psychiatric disorders) | 6 | 11
Diarrhea (Gastrointestinal disorders) | 6 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 7
Sedation (Nervous system disorders) | 5 | 8
Dizziness (Nervous system disorders) | 7 | 4
Rash (Skin and subcutaneous tissue disorders) | 2 | 8
Vomiting (Gastrointestinal disorders) | 4 | 6
Dyspepsia (Gastrointestinal disorders) | 4 | 5
Constipation (Gastrointestinal disorders) | 2 | 5
Dry Mouth (Gastrointestinal disorders) | 5 | 2
Irritability (General disorders) | 3 | 4
Pruritis (Skin and subcutaneous tissue disorders) | 4 | 3
Abdominal Pain (Gastrointestinal disorders) | 1 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Depression (Psychiatric disorders) | 2 | 3 — worse than baseline
Neck Pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Vision Blurred (Eye disorders) | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 4
Disturbance in attention (General disorders) | 1 | 3
Hypersensitivity (General disorders) | 1 | 3
Migraine (Nervous system disorders) | 3 | 1
Muscle spasm (Musculoskeletal and connective tissue disorders) | 1 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 3
Hot Flush (Endocrine disorders) | 0 | 3
Non-cardiac chest pain (Endocrine disorders) | 0 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Tinnitus (Ear and labyrinth disorders) | 3 | 0

LIMITATIONS AND CAVEATS:
Limitations of this trial include short duration of treatment (6 weeks) and generalizability due to study population composed of only females.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes